CLINICAL TRIAL: NCT07381166
Title: THE EFFECT OF METERED-DOSE INHALER TRAINING AND REMINDERS ON MEDICATION ADHERENCE IN ELDERLY INDIVIDUALS: A RANDOMIZED CONTROLLED STUDY
Brief Title: THE EFFECT OF INHALER TRAINING AND REMINDERS ON MEDICATION ADHERENCE IN ELDERLY INDIVIDUALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Sevda Ateş, Associate Professor, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-SA-01
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Elderly (People Aged 65 or More)
Keywords: elderly; Metered Dose Inhalers; reminder; adherence to treatment
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: experimental design with pre-test and post-test control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm description experimental (Experimental): The socio-demographic and descriptive characteristics, as well as questions regarding medication adherence, included in the survey form will be answered through face-to-face interviews. While the participant demonstrates how to apply the inhaler, the researcher will evaluate the participant's inhaler use according to the "Metered Dose Inhaler Skill Chart," which includes the steps for inhaler use. Each participant in the experimental group will receive metered-dose inhaler training using a demonstration method. At the end of the training, participants will be given a "Metered Dose Inhaler Use Reminder Card" and a "Metered Dose Inhaler Application Video." Participants will also receive weekly reminders via telephone. After 3 months, the experimental group will be contacted via video call to demonstrate how they use the inhaler. The researcher will evaluate the participants' medication adherence scores and record them on the survey form. If any steps are incorrectly applied, the metered
  Interventions: Other: Metered Dose Inhaler Training; Other: Metered Dose Inhaler Reminder Card; Other: Metered Dose Inhaler Application Video
- arm description control (No Intervention): The socio-demographic and demographic characteristics, as well as questions regarding medication adherence, included in the survey form will be answered through face-to-face interviews. While the participant demonstrates how to apply the inhaler, the researcher will evaluate the participant's inhaler use according to the "Metered Dose Inhaler Skill Chart," which includes the steps for inhaler use. No inhaler training or reminders will be given. Participants in the control group will be contacted by phone 3 months after the initial follow-up and asked to demonstrate how they use the inhaler. The researcher will evaluate the participants' medication adherence scores and record them on the survey form. After the data collection is complete, inhaler training will be given to the participants using a demonstration method. At the end of the training, reminder cards and a video demonstrating metered-dose inhaler application will be shared with the participants.

INTERVENTIONS:
Other: Metered Dose Inhaler Training — It is known that incorrect inhaler use is more common, especially in elderly individuals, and that common errors in metered-dose inhaler use include poor hand-mouth coordination, inability to simultaneously spray and inhale, and failure to hold the breath during inhalation. This study evaluates metered-dose inhaler use only in elderly individuals. Furthermore, not only will the inhaler application steps be evaluated, but the experimental group will also receive education and reminder interventions.
  Arms: arm description experimental
Other: Metered Dose Inhaler Reminder Card — This reminder card contains the inhaler administration steps included in the "Measured Dose Inhaler Medication Use Skill Chart". Participants in the experimental group will be able to access the medication administration steps on the reminder card before administering their inhaler medication. Participants will be asked in the final interview whether they used the reminder cards.
  Arms: arm description experimental
Other: Metered Dose Inhaler Application Video — This video was prepared by the responsible researcher, taking into account the application steps included in the "Metered Dose Inhaler Medication Use Skill Chart". Participants in the experimental group will be able to access the application steps via the inhaler video before administering their inhaler medication.
  Arms: arm description experimental

SUMMARY:
This study will evaluate the effect of metered-dose inhaler training and reminders on treatment adherence in elderly individuals.

DETAILED DESCRIPTION:
The presence of multiple comorbidities and an increased number of medications in elderly individuals are significant risk factors for non-adherence to inhaler therapy. Forgetfulness, lack of confidence in medications and difficulty understanding how to take them, depression, low self-efficacy, disease severity, and disease perception can all affect adherence to treatment. Incorrect inhaler use can lead to patients receiving insufficient medication, increased symptom burden, and negatively impact their quality of life. Furthermore, incorrect inhaler technique has been shown to increase the risk of hospitalization, emergency room visits, and the use of antibiotics and oral corticosteroids. Implementing procedures to ensure correct inhaler use is crucial in controlling critical errors in inhaler therapy. Elderly patients are more likely to have conditions such as arthritis that affect physical movement and coordination. Cognitive function also affects the ability to use inhaler devices correctly. It is known that incorrect inhaler use is more common, particularly in untrained and elderly individuals, with frequent errors including poor hand-mouth coordination, inability to synchronize spraying and inhalation, and failure to hold the breath during inhalation being common mistakes in metered-dose inhaler use. Therefore, this study will evaluate the effect of metered-dose inhaler training and reminders on treatment adherence in elderly individuals.

ELIGIBILITY:
Inclusion criteria for the study:

* Age ≥ 65 years old
* Having at least basic literacy,
* Receiving metered-dose inhaler therapy for at least 6 months,
* Being hospitalized in the pulmonary ward,
* Presenting to the pulmonary function test unit,
* Presenting to the pulmonary outpatient clinic,
* Signing the informed consent form for participation in the study,
* Having internet access and a mobile device with Android/iOS operating system,
* Being able to use a telephone,
* Having no communication barriers,
* Being able to use the inhaler without needing assistance,
* Making an error in at least one of the usage steps according to the MDI usage skills chart.

Exclusion criteria for the study:

* Age <65
* Illiteracy
* Receiving metered-dose inhaler therapy for <6 months
* Outpatient treatment
* Being hospitalized in the intensive care unit
* Being hospitalized in wards other than the pulmonary ward (such as surgery, physical therapy)
* Visiting outpatient clinics other than the pulmonary clinic (such as surgery, physical therapy)
* Not signing the informed consent form for participation in the study
* Not having internet access and a mobile device with Android/iOS operating system
* Not having telephone skills
* Having communication barriers
* Requiring assistance while using the inhaler
* Not making any errors in the usage steps according to the MDI usage skills chart
* Wanting to withdraw from the study/withdrawing from participation during the research process
* Not completing the questionnaire

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Metered Dose Inhaler Skill | the initial screening and three months after the initial screening (three months)
  The "Measured Dose Inhaler Skill Chart" involves evaluating the participant's inhaler usage and checking the application steps. Performing all steps correctly will be considered "correct inhaler technique," while performing at least one or more steps incorrectly or not at all will be considered "incorrect inhaler technique." For each step, incorrect application or omission will receive "0 points," and correct application will receive "1 point," resulting in a total score between "0 and 10." Participants who make at least "1 mistake" or score "below 10" will be included in the study. When evaluating scores based on inhaler usage steps, "0-3" points will be considered poor, "4-6" points moderate, and "7-10" points good.
Medication Adherence Reporting Scale | the initial screening and three months after the initial screening (three months)
  The scale consists of 5 items in total. The total test score is determined by summing the scores obtained from the items. Scores obtained from the scale range from 5 to 25. Higher total scores indicate better medication adherence, while lower total scores indicate poor medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Ateş, Associate Professor, Principal Investigator — Çanakkale Onsekiz Mart University
Locations (1):
- Department of Nursing, Faculty of Health Sciences, Canakkale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In the ethics committee approval and institutional permission obtained for the study, I stated that the study would not be shared anywhere other than for publication.